CLINICAL TRIAL: NCT05957003
Title: The Validity of Combined End-expiratory and End-inspiratory Occlusion Test and Tidal Volume Challenge Test for Prediction of Fluid Responsiveness in Immediate Post-cardiac Surgery Patients
Brief Title: Fluid Responsiveness in Post-cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: fluid responsiveness
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Fluid Overload; Cardiac Surgery; Postoperative Complications
MeSH Terms: conditions — Edema; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- occlusions test (Active Comparator): Combined end expiratory (EEO) and inspiratory occlusion (EIO) test. A 15-s EEO separated by a time window of 1 minute to allow the hemodynamic parameters to return to baseline followed by a 15-s EIO
  Interventions: Procedure: Combined end-expiratory occlusion and end-inspiratory occlusion test
- challenge test (Active Comparator): Tidal volume (TV) challenge test (transient increase of TV from 6 to 8 mL/kg for 1 minute)
  Interventions: Procedure: Tidal volume challenge test

INTERVENTIONS:
Procedure: Combined end-expiratory occlusion and end-inspiratory occlusion test — The EEO test will be performed by interrupting the mechanical ventilation at end-expiration over 15 seconds using the end-expiratory hold button available on the ventilator.
  The EIO test will be performed by interrupting the mechanical ventilation at end-inspiration over 15 seconds using the end-inspiratory hold button available on the ventilator.
  Arms: occlusions test
Procedure: Tidal volume challenge test — elevating tidal volume from 6 ml/kg to 8 ml/kg for only 60 seconds
  Arms: challenge test

SUMMARY:
the study aims to examine the validity of combined end-expiratory and end-inspiratory occlusion test and tidal volume challenge test for prediction of fluid responsiveness in immediate post-cardiac surgery patients

DETAILED DESCRIPTION:
multiple studies prove that dynamic variables based on heart-lung interactions accurately can predict fluid responsiveness in mechanically ventilated patients, including pulse pressure variation (PPV) and stroke volume (SV) variation.

Furthermore, passive leg raising (PLR), end-expiratory occlusion test, and tidal volume challenge test, "Mini"-fluid challenge are currently available to assess fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation
* Patients ≥18 years of age
* patients undergoing cardiac surgery (coronary artery bypass graft, valve repair/ replacement, combined cardiac surgery)
* patients with normal systolic function of the left and right ventricle
* patient is mechanically ventilated with a protective lung strategy

Exclusion Criteria:

* Patients with Spontaneously breathing activity
* Patients undergoing emergent cardiac surgery.
* Patient with severe peripheral arterial occlusive disease
* Pregnant women
* Contraindication of passive leg raising test
* unstable post-operative course
* Post-operative complications such as uncontrolled bleeding, severe neurologic impairment, or accidental mechanical complications;
* presence of residual severe tricuspid or any valvular regurgitations
* low cardiac output, low ejection fractions (EF ≤45%)
* open chest,Pao2/Fio2 ≤ 200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
The number of volume responder participants could be detected using each fluid responsiveness test | immediate postoperative period
  The number of volume responder participants could be detected using each fluid responsiveness test including tidal volume challenge test and combined end-expiratory occlusion and end-inspiratory occlusion test

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No